CLINICAL TRIAL: NCT00346034
Title: A 12 Week, Open-Label, Safety Trial Of Pregabalin In Patients With Fibromyalgia
Brief Title: This Study is An Open-Label Trial Of Pregabalin In Patients With Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0081101
Record Dates: First submitted 2006-06-28; First posted 2006-06-29 (Estimated); Results first posted 2009-03-13 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2018-11

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — 150 to 600mg/day

SUMMARY:
The main purpose of this protocol is to evaluate the long-term safety of pregabalin in patients who participated in the previous fibromyalgia Study A0081100 and who wish to receive open-label pregabalin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met the inclusion criteria for the preceding fibromyalgia Protocol A0081100, and must have received pregabalin/placebo under double-blind conditions.

Exclusion Criteria:

* Patients may not participate in the study if they experienced a serious adverse event during the previous fibromyalgia Study A0081100 which was determined to be related to the study medication by the investigator or the sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2006-12; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (46):
- Canada (11):
  - Pfizer Investigational Site, Kelowna, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Bathurst, New Brunswick
  - Pfizer Investigational Site, St. John's, Newfoundland and Labrador
  - Pfizer Investigational Site, Hawkesbury, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Drummondville, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Pointe-Claire, Quebec
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
- Denmark (2):
  - Pfizer Investigational Site, Frederiksberg
  - Pfizer Investigational Site, Svendborg
- France (5):
  - Pfizer Investigational Site, Montpellier, Cedex 5
  - Pfizer Investigational Site, Lille, Cedex
  - Pfizer Investigational Site, Clermont-Ferrand
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Saint-Priest-en-Jarez
- Germany (3):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Mannheim
  - Pfizer Investigational Site, München
- India (3):
  - Pfizer Investigational Site, Indore, Madhya Pradesh
  - Pfizer Investigational Site, Ludhiana, Punjab
  - Pfizer Investigational Site, Lucknow, Uttar Pradesh
- Italy (5):
  - Pfizer Investigational Site, Bari
  - Pfizer Investigational Site, Benevento
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Chieti Scalo
  - Pfizer Investigational Site, Pisa
- Netherlands (4):
  - Pfizer Investigational Site, Alkmaar
  - Pfizer Investigational Site, Den Helder
  - Pfizer Investigational Site, Leeuwarden
  - Pfizer Investigational Site, Zwolle
- Pfizer Investigational Site, Lisbon, Portugal
- South Korea (2):
  - Pfizer Investigational Site, Suwon, Kyeongki-do
  - Pfizer Investigational Site, Seoul
- Sweden (4):
  - Pfizer Investigational Site, Linköping
  - Pfizer Investigational Site, Mölndal
  - Pfizer Investigational Site, Örebro
  - Pfizer Investigational Site, Stockholm
- Pfizer Investigational Site, Zurich, Switzerland
- United Kingdom (5):
  - Pfizer Investigational Site, Manchester, Greater Manchester
  - Pfizer Investigational Site, Greenock, Renfrewshire
  - Pfizer Investigational Site, North Shields, Tyne and Wear
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Poole

REFERENCES:
- [Derived] Arnold LM, Emir B, Murphy TK, Zeiher BG, Pauer L, Scott G, Petersel D. Safety profile and tolerability of up to 1 year of pregabalin treatment in 3 open-label extension studies in patients with fibromyalgia. Clin Ther. 2012 May;34(5):1092-102. doi: 10.1016/j.clinthera.2012.03.003. Epub 2012 Apr 14. PMID 22503162
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081101&StudyName=This%20Study%20is%20An%20Open-Label%20Trial%20Of%20Pregabalin%20In%20Patients%20With%20Fibromyalgia%20%20%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was planned to include all eligible subjects continuing from the preceding double-blind study A0081100 NCT00333866 (Subjects had to be at least 18 years old and have met the American College of Rheumatology criteria for fibromyalgia).
Pre-assignment Details: Following the termination visit in study A0081100, subjects had an option of starting pregabalin under open-label conditions the day after the termination visit.
Groups:
- Pregabalin: Subjects began the open-label study (A0081101) medication the morning after termination visit from double-blind study (A0081100) at a fixed dose of 300 mg/day. Pregabalin daily dose was adjusted thereafter by the investigator to optimize pain control and to minimize adverse events. Adjustments to total daily doses were permitted for the remainder of the study. The minimum permissible daily dose was 150 mg/day (75 mg BID) and the maximum daily dose was 600 mg/day (300 mg BID) of pregabalin.
Period: Overall Study
Arm/Group | Pregabalin
Started | 357
Completed | 300
Not Completed | 57
Not completed — Adverse Event | 34
Not completed — Lack of Efficacy | 8
Not completed — Withdrawal by Subject | 13
Not completed — Patient Stopped Taking Study Drug | 1
Not completed — Not Willing to Follow Dosing Regimen | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pregabalin
Number analyzed (Participants) | 357
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 322
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 4 in Pain Visual Analog Scale (VAS) Score
Description: Mean Change: Observation VAS score minus Baseline score. Pain VAS: 100 mm horizontal line to rate (score) pain from 0 "no pain" to 100 "worst possible pain". Baseline = value @ double-blind screening if randomized to pregabalin during double-blind or value @ last visit from double-blind if randomized to placebo during double-blind.
Time Frame: Week 4
Population: This will include all patients who have received at least one dose of study medication and had observations at both baseline and week 4.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Pregabalin
Number analyzed (Participants) | 306
mm | -18.1 (24.1)

2. Primary Outcome: Change From Baseline to Week 12 in Pain Visual Analog Scale (VAS) Score
Description: Mean Change: Observation VAS score minus Baseline score. Pain VAS is a 100mm horizontal line used to rate (score) pain by subject from 0 "no pain" to 100 "worst possible pain". Baseline=value @ double-blind screening if randomized to pregabalin during double-blind OR value @ last visit from double-blind if randomized to placebo during double-blind.
Time Frame: Week 12 (end of treatment)
Population: This will include all patients who have received at least one dose of study medication and observations at both baseline and week 12.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Pregabalin
Number analyzed (Participants) | 335
mm | -20.1 (26.8)

ADVERSE EVENTS:
Arm/Group | Pregabalin
Serious Adverse Events (participants affected / at risk) | 6
Other Adverse Events (participants affected / at risk) | 173
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Pregabalin
Diarrhea (Gastrointestinal disorders) | 1/357
Melaena (Gastrointestinal disorders) | 1/357
Vomiting (Gastrointestinal disorders) | 1/357
Urinary tract infection (Infections and infestations) | 1/357
Fall (Injury, poisoning and procedural complications) | 1/357
Wrist fracture (Injury, poisoning and procedural complications) | 1/357
Spinal osteoarthritis (Injury, poisoning and procedural complications) | 1/357
Myoclonus (Nervous system disorders) | 1/357
Vulva cyst (Reproductive system and breast disorders) | 1/357
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1/357
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Pregabalin
Dizziness (Nervous system disorders) | 85/357
Headache (Nervous system disorders) | 33/357
Somnolence (Nervous system disorders) | 30/357
Vertigo (Ear and labyrinth disorders) | 12/357
Constipation (Gastrointestinal disorders) | 15/357
Dry mouth (Gastrointestinal disorders) | 14/357
Nausea (Gastrointestinal disorders) | 21/357
Vomiting (Gastrointestinal disorders) | 13/357
Fatigue (General disorders) | 24/357
Oedema peripheral (General disorders) | 12/357
Nasopharyngitis (Infections and infestations) | 11/357
Weight increased (Investigations) | 14/357

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 mo from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results